CLINICAL TRIAL: NCT02934698
Title: An Efficacy and Safety Study of Ivacaftor in Patients With Cystic Fibrosis and Two Splicing Mutations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00052526
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ivacaftor (Experimental): There is only one arm to this study. The two sisters with Cystic Fibrosis will both receive Ivacaftor for 6 months for their treatment.
  Interventions: Drug: Ivacaftor

INTERVENTIONS:
Drug: Ivacaftor — Subjects will be treated with ivacaftor for 6 months and followed for 7 months and will undergo assessments along the way to measure sweat chloride and sputum amounts.

SUMMARY:
This postmarketing N of 2 study is designed to evaluate the efficacy and safety of open-label ivacaftor treatment in two sisters with cystic fibrosis and pancreatic sufficiency.

DETAILED DESCRIPTION:
The two sisters have a splicing mutation that is predicted to respond favorably to ivacaftor therapy. In addition to measurement of usual clinical outcomes (i.e. lung function, nutritional status), there is great interest on the impact on nontuberculous mycobacteria (NTM) airways infection.

Subjects will undergo sputum cultures at baseline and monthly during treatment, initially in the absence of anti-NTM therapy but with the intent to treat with antibiotics if there is persistence of the infection in cultures. Other clinical outcomes will include changes in sweat chloride, lung function and weight. Safety measures will include periodic assessment of liver enzymes. All serious and non-serious adverse events will be collected

ELIGIBILITY:
Inclusion Criteria:

* Subjects are >18 years of age and able to provide informed consent.
* Subjects reside in the US and are willing to be treated with ivacaftor.
* Subjects have the splicing mutation of interest.
* Subjects are willing and able to perform requirements of the study.

Exclusion Criteria:

* There are no relevant exclusion criteria for this n-of-2 study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Flume, MD, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ivacaftor
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ivacaftor
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 37 [36 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume
Description: Absolute change in percent predicted in 1 second FEV1 from baseline through week 24
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: percentage of predicted
Arm/Group | Ivacaftor
Number analyzed (Participants) | 2
percentage of predicted | 4 [3 to 5]

2. Secondary Outcome: Sputum Results
Description: Achievement of mycobacterial culture conversion (negative culture)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ivacaftor
Number analyzed (Participants) | 2
Participants | 2

3. Secondary Outcome: Sweat Chloride
Description: Testing efficacy through gathering absolute change in sweat chloride from baseline through week 24
Time Frame: 24 Weeks
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Ivacaftor
Number analyzed (Participants) | 2
mmol/L | -5.7 [-8 to -3.5]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Ivacaftor
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivacaftor (N=2)
Sinus congestion (Infections and infestations) | 2 (4)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) — Nose
palpitations (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT02934698/Prot_SAP_000.pdf